CLINICAL TRIAL: NCT05578911
Title: Medical Follow-up and Self-medication Among Medical Students
Acronym: AutoMed-Int
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_005_AutoMed-Int
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Medical Student
Keywords: medical student; medical follow-up; self medication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: "medical students" group — medical student in general practice or in specialty medicine

SUMMARY:
As health actors, medical students educate patients to have regular medical follow-up and give them justified medical prescriptions. Regarding their own health, medical students do not seem to apply these same principles.

The medical follow-up of medical students seems insufficient, which can be explained by the lack of medical follow-up by occupational medicine, a consequent work time, but also the fear of judgment by colleagues Moreover, medical student have an easy access to all types of prescriptions and therefore the ease of self-prescription and self-medication. Medical students may also overestimate their medical knowledge and may not be objective about their symptomatology.

DETAILED DESCRIPTION:
The aim of the study will be to describe medical follow-up and self-medication among medical students

ELIGIBILITY:
Inclusion Criteria:

* medical student in general practice or in specialty medicine
* agreeing to participate in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: medical student in general practice or in specialty medicine
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
self-medication | Day 0
  Number of medical students with prescription for themself of a medical treatment

SECONDARY OUTCOMES:
self-prescription | Day 0
  Number of medical students with prescription for themself of an biological analysis and/or a medical imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Ufr Medecine Urca, Reims, France